CLINICAL TRIAL: NCT03444207
Title: Effect of Endurance and Endurance-Strength Training on Inflammatory Markers in Women With Abdominal Obesity
Acronym: ENDOFIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Pawel Bogdanski, Professor, Poznan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1077/12; 753/13
Record Dates: First submitted 2018-02-13; First posted 2018-02-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Obesity
Keywords: obesity; inflammation; C-reactive protein; training; tumor necrosis factor alfa
MeSH Terms: conditions — Obesity; Inflammation | interventions — Endurance Training

STUDY DESIGN:
Intervention Model Description: The study was designed as a prospective randomized trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Endurance training
  Interventions: Behavioral: Endurance training
- Group B (Experimental): Endurance-strength training
  Interventions: Behavioral: Endurance-strength training

INTERVENTIONS:
Behavioral: Endurance training — The women in group A underwent endurance exercise on cycle ergometers (Schwinn Evolution, Schwinn Bicycle Company, Boulder, Colorado, USA). Exercise sessions consisted of a five-minute warm-up (stretching exercise) at low intensity (50%-60% of maximum heart rate), a 45-minute exercise (at 50%-80% of maximum heart rate), five minutes of cycling without a load, and five minutes of closing stretching and breathing exercise of low intensity.
  Arms: Group A
Behavioral: Endurance-strength training — Group B performed endurance-strength exercise consisting of a five-minute warm-up (stretching exercises) of low intensity (50%-60% of maximum heart rate), a strength component, an endurance component, 5 minutes cycling without a load, and a 5 minutes closing stretching and breathing exercise of low intensity. The 20-minute-long strength component was performed using a neck barbell and a gymnastic ball. Directly after the strength exercise, the women took part in a 25-minute endurance exercise on cycle ergometers (Schwinn Evolution, Schwinn Bicycle Company, Boulder, Colorado, USA) at 50%-80% of maximum heart rate.
  Arms: Group B

SUMMARY:
The aim of this study was to compare the effects of three months' endurance training and three months' endurance-strength training on inflammatory markers in women with abdominal obesity.

DETAILED DESCRIPTION:
Study patients. Written informed consent was obtained from all subjects. The study meets the standards of the Declaration of Helsinki in its revised version of 1975 and its amendments of 1983, 1989, and 1996.

Study design. The study was designed as a prospective randomized trial. Subjects were randomly divided into two groups, A and B, using a randomization list. Both groups performed three month of physical training. Group A underwent endurance training, while group B performed endurance-strength training. Aside from the training, all subjects were instructed to maintain the physical activity and diet that they had been practicing so far. At baseline and after three months of physical training, blood samples for laboratory analyses were taken, anthropometric measurements were performed for both groups.

Intervention. The exercise program lasted three months, with three sessions per week. Women in both groups participated in a total of 36 training sessions. The women in group A underwent endurance exercise on cycle ergometers (Schwinn Evolution, Schwinn Bicycle Company, Boulder, Colorado, USA). Exercise sessions consisted of a five-minute warm-up (stretching exercise) at low intensity (50%-60% of maximum heart rate), a 45-minute exercise (at 50%-80% of maximum heart rate), five minutes of cycling without a load, and five minutes of closing stretching and breathing exercise of low intensity. Group B performed endurance-strength exercise consisting of a five-minute warm-up (stretching exercises) of low intensity (50%-60% of maximum heart rate), a strength component, an endurance component, 5 minutes cycling without a load, and a 5 minutes closing stretching and breathing exercise of low intensity. The 20-minute-long strength component was performed using a neck barbell and a gymnastic ball. Directly after the strength exercise, the women took part in a 25-minute endurance exercise on cycle ergometers (Schwinn Evolution, Schwinn Bicycle Company, Boulder, Colorado, USA) at 50%-80% of maximum heart rate. Both the endurance and endurance-strength training were comparable in exercise volume; the only difference was the nature of the effort.

ELIGIBILITY:
Inclusion Criteria:

* informed written consent;
* simple obesity;
* age from 18 to 65 years;
* body fat content, assessed by electrical bioimpedance, equal to or more than 33%;
* waist circumference more than 80 cm;
* stable body weight in the one month prior to the trial.

Exclusion Criteria:

* secondary form of excess body mass
* secondary form of arterial hypertension
* mean systolic blood pressure > 140 mmHg and/or mean diastolic blood pressure > 90 mmHg;
* diabetes;
* ischemic heart disease;
* stroke;
* heart failure;
* history of malignancy;
* clinically significant heart arrhythmias;
* a history of use of any dietary supplement;
* serious liver or kidney damage;
* abnormal thyroid gland function;
* clinically significant inflammation, connective tissue disease, or arthritis;
* nicotine, alcohol, or narcotic abuse;
* infection;
* pregnancy, childbirth, or lactation;
* any other condition that would make participation not in the best interest of the subject, or could prevent the efficacy of the study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-representation of gender identity.
Enrollment: 38 (Actual)
Dates: Start 2012-12-06 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
C-reactive protein (CRP) at baseline | At baseline
  Serum concentration of C-reactive protein at baseline
CRP after three months of physical training | after three months of physical training
  Serum concentration of C-reactive protein after three months of physical training

SECONDARY OUTCOMES:
tumor necrosis factor alpha (TNFα) at baseline | at baseline
  Serum concentration of tumor necrosis factor alpha at baseline
TNFα after three months of physical training | after three months of physical training
  Serum concentration of tumor necrosis factor alpha after three months of physical training
soluble receptor 2 of TNF alpha (sTNF R2) at baseline | At baseline
  Serum concentration of soluble receptor 2 of TNF alpha at baseline
sTNF R2 after three months of physical training | after three months of physical training
  Serum concentration of soluble receptor 2 of TNF alpha after three months of physical training
interleukin 6 (IL-6) at baseline | At baseline
  Serum concentration of interleukin 6 at baseline
IL-6 after three months of physical training | after three months of physical training
  Serum concentration of interleukin 6 after three months of physical training
interleukin 1 (IL-1) at baseline | At baseline
  Serum concentration of interleukin 1 at baseline
IL-1 after three months of physical training | after three months of physical training
  Serum concentration of interleukin 1 after three months of physical training
visfatin at baseline | At baseline
  Serum concentration of visfatin at baseline
visfatin after three months of physical training | after three months of physical training
  Serum concentration of visfatin after three months of physical training
Body mass at baseline | At baseline
  Body mass at baseline
Body mass after three months of physical training | after three months of physical training
  Body mass after three months of physical training
Body height at baseline | At baseline
  Body height at baseline
Body height after three months of physical training | after three months of physical training
  Body height after three months of physical training

CONTACTS AND LOCATIONS:
Overall Officials: Pawel Bogdanski, Prof., Study Chair — Department of Education and Obesity Treatment and Metabolic Disorders; Poznan University of Medical Sciences
Locations (1):
- Department of Education and Obesity Treatment and Metabolic Disorders; Poznan University of Medical Sciences, Poznan, Poland

REFERENCES:
- [Derived] Jamka M, Piotrowska-Brudnicka SE, Karolkiewicz J, Skrypnik D, Bogdanski P, Cielecka-Piontek J, Sultanova G, Walkowiak J, Madry E. The Effect of Endurance and Endurance-Strength Training on Bone Health and Body Composition in Centrally Obese Women-A Randomised Pilot Trial. Healthcare (Basel). 2022 Apr 28;10(5):821. doi: 10.3390/healthcare10050821. PMID 35627958